CLINICAL TRIAL: NCT02733068
Title: A Phase III Double Blinded, Randomized Controlled Study to Evaluate Efficacy of Protection Against HPV-16 and 18 Related Diseases, Immunogenicity and Safety of HPV-16/18 Vaccine in Healthy Females Aged 18-30 Years
Brief Title: A Phase III Study of Human Papillomavirus (HPV)-16/18 Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 311-HPV-1003
Record Dates: First submitted 2016-02-19; First posted 2016-04-11 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV-16/18 vaccine (Experimental): Including 6000 participants who received the HPV-16/18 vaccine 0.5ml.
  Interventions: Biological: HPV-16/18 vaccine
- HPV-16/18 placebo (Placebo Comparator): Including 6000 participants who received the HPV-16/18 placebo 0.5ml.
  Interventions: Biological: HPV-16/18 placebo

INTERVENTIONS:
Biological: HPV-16/18 vaccine — 0.5ml of recombinant human papillomavirus virus-like particle vaccine (Type 16 and 18 L1 Proteins, Yeast) on upper arm deltoid muscle with a three-dose-schedule (0, 2, 6 months).
  Arms: HPV-16/18 vaccine
Biological: HPV-16/18 placebo — 0.5ml of placebo on upper arm deltoid muscle with a three-dose-schedule (0, 2, 6 months).
  Arms: HPV-16/18 placebo

SUMMARY:
A Phase III Double Blinded, Randomized Controlled Study to Evaluate Efficacy of Protection Against HPV-16 and 18 Related Diseases, Immunogenicity and Safety of Recombinant Human Papillomavirus Virus-like Particle Vaccine (Type 16 and 18 L1 Proteins, Yeast) in Healthy Females Aged 18-30 Years.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, double blinded, placebo controlled study. The study vaccine is recombinant human papillomavirus bivalent (types 16 and 18) vaccine (Yeast), the placebo is aluminium phosphate diluent.

This study planned to enrol 12000 healthy female aged 18-30 in 10 study sites. Each participants will received a three-dose schedule of vaccine or placebo randomly but with the proportion controlled as 1:1 for vaccine group and placebo group. After each inoculation, the immediate reaction will be observed for 30 minutes, and the local and systemic reaction will be systematically observed for 7 days. After the first inoculation, adverse event will be collected until one month after the final inoculation, while serious adverse event will be collected until 6 months after the final inoculation. Blood samples will be collected before the first inoculation, and one month after the final injection, blood samples will also be collected in a group of participants containing 800 people to detect antibody titer.

Follow-up visit will be conducted 14 times: month 0, month 0 + 8 days, month 2, month 2 + 8 days, month 6, month 6 + 8 days, month 7, month 12, month 18, month 24, month 30, month 36, month 48, month 60. When cervical intraepithelial neoplasia grade 2+ (CIN2+) is indicated, the participant will receive standard treatment and drop out from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 healthy female
* enable to provide an legal identification
* have the ability to understand and sign the Informed Consent Form
* confirmed by the investigator that the participant has the ability to comply with the protocol requirements
* agreed to use effective contraceptive method in 7 months or has no plan of pregnancy
* can avoid vaginal sex within two days (48 hours) before every interview; don't employ a vaginal douche or any other intervention which can influence the gynecological examination and sample collection

Exclusion Criteria:

* has received HPV vaccine previously; have received other research or unregistered product (drug or vaccine) within 30 days before the first injection
* within three months before the first injection, has had received a whole-blood, plasma or immunoglobulin treatment, or planed to receive such treatments during the research period; within 28 days before the research, has had received attenuated live vaccine; or within 14 days has had received inactivated vaccine
* has a history of allergic reaction which requires medical intervention; has allergic reaction for vaccine or vaccine-containing elements; has serious adverse effect history for vaccine
* has a history of epilepsy, convulsion or has a family history of mental diseases
* has immunodeficiency diseases including: AIDS, HIV infection, lymphoma, leukemia, Systemic Lupus Erythematosus, rheumatoid arthritis, Juvenile Rheumatoid Arthritis, inflammatory bowel disease
* used immunosuppressor for treatment or corticosteroid drugs for systemic medication in 6 months
* asplenia, functional asplenia, or splenectomize
* liver and kidney diseases, serious cardiovascular diseases, diabetes, history of malignant tumor
* coagulation disorders
* in menstrual period or acute diseases
* pregnant, or less than 8 weeks after delivery
* has a history of sexual transmitted disease
* had total hysterectomy or pelvic radiotherapy
* has cervical abnormalities
* abnormal screening results for cervical cancer or had CIN in two years
* according to the judgement of investigator, participant has conditions that were not suitable for this trial
* planning to move out of the clinical trial site during the research period
* never has vaginal sexual activity

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12000 (Actual)
Dates: Start 2014-11-02; Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Cervical intraepithelial neoplasia grade 2 or more (CIN 2+) caused by HPV type 16 and/or 18. | five years
  Among the 14 follow-up visits which will be conducted during the study, 9 visits are gynecological follow-up visits. In these gynecological visits, cervical samples will be collected to conduct HPV DNA detection and cytological detection to evaluate whether occurred cervical intraepithelial neoplasia (CIN) and what grade of neoplasia occurred.

SECONDARY OUTCOMES:
Persistent infection of HPV type 16 and/or 18. | one year
  Two continuously visits with a interval of 6 months indicate the same type of HPV infection can be regard as persistent infection.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Principal Investigator — Guangxi Center for Disease Prevention and Control(GXCDC)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi L, Gao X, Huang L, Gao Z, Li J, Yu B, Fan H, Li G, Wang Y, Li Q, Yuan L, Li C, Mo Z; HPV1003 Study group. Efficacy, safety and immunogenicity of a recombinant human papillomavirus bivalent (types 16, 18) vaccine in healthy 18-30-year-old Chinese women: a phase III, double-blind, randomized, controlled trial. BMC Infect Dis. 2025 Dec 18. doi: 10.1186/s12879-025-12064-1. Online ahead of print. PMID 41413453